CLINICAL TRIAL: NCT04254744
Title: Systemic Inflammatory Response Syndrome Cyanotic and Acyanotic Children Undergoing Cardiac Surgery
Brief Title: SIRS in Cyanotic and Acyanotic Children in Cardiac Surgery
Acronym: SIRS
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Feride Karacaer, Associated professor, Cukurova University
Other Study IDs: SIRS, cardiac surgery
Record Dates: First submitted 2019-10-28; First posted 2020-02-05 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: SIRS; Pediatric Cardiac Surgery
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Acyanotic children: Acyanotic children undergoing cardiac surgery due to congenital heart disease
  Interventions: Drug: Sevoflurane
- Cyanotic children: Cyanotic children undergoing cardiac surgery due to congenital heart disease
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane inhalation for anesthesia

SUMMARY:
Systemic inflammatory response syndrome (SIRS) is frequently observed in children after open-heart surgery and has been associated with both cardiopulmonary bypass and surgical trauma. Children with congenital cyanotic heart disease (CCHD) have complex changes in all blood values and clotting profiles due to chronic hypoxemia. Increased erythrocyte count decreases plasma and coagulation factors, platelet count and function. Therefore, blood and blood products transfusion may increase during intraoperative and postoperative periods. In addition, durations of cardiopulmonary bypass may prolong due to the complex defects of children with CCHD. The aim of this study is to investigate postoperative SIRS rates and risk factors in cyanotic and acyanotic children undergoing open heart surgery for congenital heart disease.

DETAILED DESCRIPTION:
Systemic inflammatory response syndrome (SIRS) in adults has been defined as a non-specific systemic inflammatory process in the absence of infection, following incidents such as trauma, burns, pancreatitis, or major surgery. For children, age-specific SIRS criteria were established by the International Pediatric Sepsis Consensus Conference in 2005. SIRS was defined as presence of at least two out of four parameters, one of which must be an abnormal temperature or leukocyte count. The two other criteria consist of either an elevated heart rate or respiratory rate. SIRS is frequently observed in children after open-heart surgery and has been associated with both cardiopulmonary bypass and surgical trauma. Following cardiac surgery the pathophysiological mechanisms of SIRS involve a cytokine-mediated general capillary leakage followed by intravascular volume depletion, generalized edema, circulatory compromise, and altered microcirculation. The inflammatory process may further impair the function of the lung, myocardium, kidney, liver, intestine, and brain.

Children with congenital cyanotic heart disease (CCHD) have complex changes in all blood values and clotting profiles due to chronic hypoxemia. Increased erythrocyte count decreases plasma and coagulation factors, platelet count and function. Therefore, blood and blood products transfusion may increase during intraoperative and postoperative periods. In addition, durations of cardiopulmonary bypass may prolong due to the complex defects of children with CCHD. Previous studies have reported that the duration of CPB and the amount of fresh frozen plasma transfusion increase SIRS formation.

The aim of this study is to investigate postoperative SIRS rates and risk factors in cyanotic and acyanotic children undergoing open heart surgery for congenital heart disease.

Patients aged between 0-16 years and undergoing open heart surgery for cyanotic and acyanotic congenital heart disease will be included in the study. Patients with preoperative renal failure or hepatic disease will be excluded. Patient's age, weight, comorbidities, details of previous operation will be recorded. Preoperative hematocrit value, white blood cell and platelet counts, biochemical parameters (blood urea nitrogen, creatinine, electrolyte values), diagnosis of CCHD, RACHS1 (risk adjustment for surgery for congenital heart disease) will be recorded. In intraoperative period; operation time, CPB time, aortic cross-clamp time, circulatory arrest time, body temperature and lowest body temperature reached during CPB, cardioplegia amount, The ACT (activated coagulation time), urine amount will be recorded. Intraoperative blood gas values, lactate, mean arterial pressure, glucose values will be recorded at 30 min intervals. The amount of crystalloid and colloid, erythrocyte, fresh frozen plasma, platelet and cryoprecipitate used in intraoperative period will be recorded. Heparin and protamine doses administered will be recorded. Vasoactive agents (dopamine, dobutamine, adrenaline, nitroglycerine) used in intraoperative period will be recorded.

During the postoperative intensive care period; arterial blood gases and lactate, hematocrit, liquid (crystalloid and colloid) and blood products administered will be monitored at 6th, 24th and 48th hours. The vasoactive agents used, the inotropic score, the amount of urine and the use of diuretics will be recorded. Length of stay ICU, duration of mechanical ventilation, length of stay hospital will be recorded.

Diagnosis of SIRS; in the postoperative period, the age-specific SIRS criteria determined by the International Pediatric Sepsis Consensus Conference will be used. Patients will be evaluated for the diagnosis of SIRS at postoperative 6th, 12th, 24th and 48th hours. SIRS rates and risk factors in cyanotic and acyanotic patients will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 0-16 years
* undergoing open heart surgery for cyanotic and acyanotic congenital heart disease

Exclusion Criteria:

* Patients with preoperative renal failure
* Patients with preoperative hepatic disease
* Patients with preoperative inflammatory disease
* Patients using anti-inflammatory drug

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with congenital heart disease
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
White blood cell count | 48 hours after arrival in Intensive care unit
body temperature | 48 hours after arrival in Intensive care unit
heart rate | 48 hours after arrival in Intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No